CLINICAL TRIAL: NCT07359729
Title: "Deep Breathing Is More Effective Than Virtual Reality in Reducing Venipuncture Pain in Adults, With Comparable Effects on Anxiety: A Randomized Controlled Trial"
Brief Title: Deep Breathing and Virtual Reality for Venipuncture Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma del Estado de Hidalgo (Other)
Responsible Party: Principal Investigator, Mario Isidoro Ortiz Ramírez, Doctor of Science specializing in Pharmacology, Universidad Autónoma del Estado de Hidalgo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Folio: "232"/2024
Record Dates: First submitted 2025-11-25; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Anxiety; Virtual Reality; Breathing Exercises; Pain Measurement; Patient Satisfaction
Keywords: Acute pain; Pain management; Physiological parameters; Venipuncture; Procedure anxiety
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Patient Satisfaction; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (VR) (Experimental): Type of intervention: Device (VR glasses) Description: Wearing virtual reality glasses with immersive video "Dali's Dreams" for 5 minutes
  Interventions: Device: Virtual reality viewer
- Deep Breathing (RP) (Experimental): Type of intervention: Procedure Description: Diaphragmatic deep breathing technique synchronized with venipuncture
  Interventions: Behavioral: Conscious breathing
- Control Group (CG) (No Intervention): Standard venipuncture procedure without additional intervention

INTERVENTIONS:
Device: Virtual reality viewer — Participants wore virtual reality headsets with the immersive video 'Dalí's Dreams,' a 360° audiovisual experience based on the surrealist work of Salvador Dalí, lasting 5 minutes. The viewing began immediately before the venipuncture and continued throughout the procedure.
  Arms: Virtual Reality (VR)
Behavioral: Conscious breathing — "Participants were instructed and supervised in a deep diaphragmatic breathing technique that consisted of: 1) Maximum nasal inhalation, 2) Holding the breath for 5-10 seconds, and 3) Controlled and complete exhalation. Breathing was performed in sync with the moment of venipuncture."
  Arms: Deep Breathing (RP)

SUMMARY:
This study will evaluate the efficacy of two non-pharmacological techniques-virtual reality (VR) and deep breathing (DB)-in reducing pain and anxiety during venipuncture in adults. A total of 264 participants will be randomly assigned to use VR, practice DB, or receive the standard procedure (control group). Pain intensity will be measured using a Visual Analog Scale (VAS) immediately after venipuncture. Anxiety will be assessed using a VAS for anxiety and the 6-item State-Trait Anxiety Inventory (STAI-6). Physiological parameters (blood pressure and heart rate) will also be recorded. The study aims to determine which technique is more effective for pain and anxiety reduction, and to assess participant satisfaction and safety.

DETAILED DESCRIPTION:
Objective To evaluate and compare the efficacy of virtual reality (VR) and deep breathing (DB) as non-pharmacological techniques for reducing pain and anxiety during venipuncture in adult participants.

Background Venipuncture is one of the most frequent medical procedures and a significant source of pain and anticipatory anxiety for patients. While non-pharmacological interventions such as virtual reality and deep breathing have shown positive results in previous studies, comparative evidence of their efficacy in adult populations, particularly in Latin American contexts, remains scarce.

Methods This is a randomized controlled trial with three parallel groups. A total of 264 adult participants will be randomly assigned to: 1) VR group (n=72), 2) DB group (n=76), or 3) Control group (n=116). The intervention will be administered during the venipuncture procedure. Pain intensity will be measured using a Visual Analog Scale (VAS) immediately after venipuncture. Anxiety will be assessed using both a VAS for anxiety and the 6-item State-Trait Anxiety Inventory (STAI-6) before and after the procedure. Physiological parameters (blood pressure and heart rate) will be recorded at rest and immediately after venipuncture. Data will be analyzed using Analysis of Covariance (ANCOVA) adjusted for age and non-parametric tests as appropriate.

Outcomes The primary outcome is pain intensity during venipuncture. Secondary outcomes include anxiety levels, physiological parameters, and participant satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65
* With the cognitive capacity to answer questionnaires
* Requiring venipuncture in the forearm
* Who agreed to participate voluntarily

Exclusion Criteria:

* Intolerance to virtual reality
* Uncorrectable visual or hearing impairments
* Alcohol or illegal drug use within the previous 12 hours
* Heart disease
* Chronic use of analgesics or anticoagulants
* Skin conditions at the puncture site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Pain Intensity During Venipuncture | Immediately post-venipuncture (within the first 2 minutes after the procedure)
  Pain intensity measured using a Visual Analog Scale (VAS), scored from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable". Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Procedure-related anxiety (VAS-A) | Before procedure (pre-venipuncture) and immediately after procedure (within 2 minutes post-venipuncture)
  Anxiety measured using Visual Analog Scale for Anxiety (VAS-A), scored from 0 to 10, where 0 = "no anxiety" and 10 = "worst anxiety imaginable". Higher scores indicate greater anxiety.
Procedure-related anxiety (STAI-6) | Before procedure (pre-venipuncture) and immediately after procedure (within 2 minutes post-venipuncture)
  Anxiety measured using 6-item State-Trait Anxiety Inventory (STAI-6), scored from 6 to 24 points. Higher scores indicate greater state anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela de Medicina UAEH Campus Ramirez Ulloa, Pachuca, Hidalgo, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared to protect patient confidentiality and privacy, in accordance with local data protection regulations and the guidelines of the ethics committee that approved the study. Aggregated information and study results will be made available through scientific publication.